CLINICAL TRIAL: NCT07105410
Title: The Influence of Nociception on Exercise Induced Fatigue: the Analgesic Role of Acute Exercise and Long-term Training of Different Exercise Modalities
Brief Title: Hypoalgesic Effects of Exercise and Training of Different Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Principal Investigator, André Dias Gonçalves, MSc, Faculdade de Motricidade Humana
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CEIFMH Nº33/2021
Record Dates: First submitted 2025-07-17; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Training; Exercise; Fatigue; Occlusion
Keywords: hypoalgesia; pain
MeSH Terms: conditions — Motor Activity; Fatigue; Bites and Stings; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PECO and No-PECO (Experimental)
  Interventions: Other: Aim #1: The effect of post-exercise circulatory occlusion on H-reflex and V-wave
- Aerobic, Anaerobic and Dynamic Resistance Exercise (Experimental)
  Interventions: Other: Aim #2: The hypoalgesic effects of acute exercise of different modalities
- Aerobic, Anaerobic, Dynamic Resistance Training and Control Group (Experimental)
  Interventions: Other: Aim #3: The hypoalgesic effects of chronic training of different modalities

INTERVENTIONS:
Other: Aim #1: The effect of post-exercise circulatory occlusion on H-reflex and V-wave — Aim #1 follows a randomized and crossover design in which 16 young and healthy males are evaluated during thigh circulatory occlusion performed after a submaximal isometric plantar flexion contraction (PECO day). In the other session, participants are evaluated during free-flow conditions and without previous fatiguing contraction (no-PECO day). In PECO day, participants complete a 3-min contraction at 40% of maximal force. Then, for testing, blood flow from lower-leg is blocked during 4 min, by an inflatable cuff around the ipsilateral thigh before task termination, during which H- reflex is tested. At the end of recordings, the cuff is deflated. Participants ware allowed to rest for 5-10 min. Then, they are requested to perform a new 3 min contraction with the cuff being inflated before task termination. The cuff remains inflated for ~ 2 min during which V-wave recordings are obtained. In both days, leg pain intensity is reported by participants and brachial AP is measured.
  Arms: PECO and No-PECO
Other: Aim #2: The hypoalgesic effects of acute exercise of different modalities — Aim #2 follows a randomized and crossover-controlled design, consisting on two experimental sessions. 24 healthy male (all diferent from Experiment 1) are randomly allocated to one of the following exercising regimens: aerobic, anaerobic or dynamic resistance (8 participants for each exercise group). In one of the experimental days, participants are evaluated for pain sensitivity and neuromuscular responses both before and after a lower-limb acute exercise protocol (exercise day) and in the other day before and after 15 min of quiet rest (non-exercise day). In both sessions, participants are evaluated for rectus femoris, upper trapezius and biceps brachiis muscles pressure pain threshold, followed by the application of a cold pain tolerance test on the foot. The intensity of pain is reported by a 0-100mm VAS and AP and HRV continously measured. Then, participants are tested for H-reflex and V-wave excitability during PECO, with leg pain intensity (0-10) and brachial AP recorded.
  Arms: Aerobic, Anaerobic and Dynamic Resistance Exercise
Other: Aim #3: The hypoalgesic effects of chronic training of different modalities — Aim #3 follows a randomized-controlled design. 32 healthy male (all the 24 participants from Experimental 2 plus 8 new subjects) are randomly allocated to one of the following groups: aerobic, anaerobic, dynamic resistance training and no-training (control) (8 participants for each group). Each intervention group perform 6 weeks of exercise training (3x week). Participants allocated to each training group are evaluated before and after training (2 assessment days in each time-point). On one day participants are tested for pressure pain threshold and cold pain tolerance with concomitant measures of pain ratings (0-100mm VAS), AP and HRV. The influence of metaboreflex activation on H-reflex and V-wave is also measured (during PECO). In addition, during PECO ischemic pain rating and AP are obtained. On another day, participants are evaluated for motor performance (maximal oxygen uptake, maximal voluntary contraction and peak power) and neuromuscular adaptations (i.e. H-reflex and V-wave)
  Arms: Aerobic, Anaerobic, Dynamic Resistance Training and Control Group

SUMMARY:
Further research is needed to explore the analgesic effects of post-acute and chronic exercise and if effects are partially dependent on lower H-reflex/V-wave inhibition by group III and IV muscle afferents desensitization. In addition, it is important to note that the available research examining the interaction between exercise (acute and chronic) and pain did not compare the effect of different exercise modalities. Moreover, since discharge rate of III and IV afferents is highly dependent on specific task-metabolic requirements, it is relevant to determine if exercise modality differentially modulates the possible analgesic response via metaboreflex desensitization.

Therefore, with this project, the investigators aim at exploring the influence of experimentally induced metaboreflex activation (group III and IV afferents) (maintained submaximal isometric contraction followed by blood-flow occlusion - post-exercise circulatory occlusion (PECO)) Vs. a control condition (no isometric contraction nor blood flow occlusion), on H-reflex recruitment curve and V-wave excitability (aim #1). Since the activation of group III/IV afferents can inhibit the corticospinal pathway, the investigators hypothesize that the normalized maximal amplitude of H- and V-wave and the slope of the ascending limb of the H-recruitment curve will decrease with metaboreflex activation (during PECO). Additionally, the investigators intend to examine the acute impact of different lower-limb exercise regimens (aerobic, anaerobic and dynamic resistance) on pain sensitivity (by the application of a foot cold pain tolerance test, by determining pressure pain threshold of exercising and non-exercising muscles and through self-reported leg ischemic pain ratings (0-10 Cook scale) - during PECO) (aim #2). Participants are also asked to mark the intensity of cold pain sensation using a visual analogue scale (VAS) with a horizontal line of 100mm, every 30 s of testing.This will allow the investigators to investigate the analgesic role of different acute exercise paradigms through possible metaboreflex desensitization given by altered neuromuscular responses at post-exercise time point (attenuated inhibition of H-reflex and V-wave amplitude during PECO). Also, once past research has shown that muscle metaboreflex activation reduces the sensitivity of the baroreflex, the investigators will measure arterial pressure (AP) and heart rate variability (HRV) during cold test and AP during ischemic testing. Despite all exercise modalities could enhance reducing pain sensibility after exercise, the investigators hypothesize that resistance and anaerobic exercise stimuli will enhance pain threshold/tolerance and reduced pain ratings via metaboreflex desensitization compared to that seen with endurance exercise (attenuated increase of AP and sympathetic component of HRV during cold pressor test and attenuated increase of AP during ischemic pain test). Finally, the investigators intend to explore the impact of long-term aerobic, anaerobic and resistance training on pain sensibility, using the same tests of aim #2 (aim #3). The investigators hypothesize that chronic EIH will be of greater magnitude after anaerobic and resistance exercise training vs. endurance training. This will be related with attenuated inhibition of H-reflex and V-wave amplitude measured during PECO and attenuated increase of AP and sympathetic component of HRV during metaboreflex activation after those training modalities. Nevertheless, the investigators expect to see an increased motor performance in all training regimens via heightened H-reflex (aerobic and anaerobic groups) and V-wave (resistance group) excitability.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 35 years males
* Healthy (health status determined from a health-screening questionnaire performed at study admission)
* Normal arterial blood pressure (ABP) (cut-off values for systolic arterial pressure (SAP) and diastolic arterial pressure (DAP) of ≤ 120/80 mmHg)

Exclusion Criteria:

* Neurologic disease
* Metabolic disease
* Cardiovascular disease
* Respiratory disease
* Musculoskeletal issues in the 3 previous months limiting exercise performance
* Taking any chronic medications for the treatment of pain or had any pain related condition

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
H-reflex | During PECO and No-PECO conditions (aim #1); Pre-post acute exercise during PECO (aim #2); Pre-post 6 weeks of training during PECO (aim #3)
  With soleus electromyographic recording electrode (Delsys) and electrical stimulation of the tibial nerve (Stimsola) the H-reflex recruitment curve parameters (spinal excitability) will be obtained in a 4-min protocol
V-wave | During PECO and No-PECO conditions (aim #1); Pre-post acute exercise during PECO (aim #2); Pre-post 6 weeks of training during PECO (aim #3)
  With soleus electromyographic recording electrode (Delsys) and electrical stimulation of the tibial nerve (Stimsola) the V-wave parameters (spinal and supraspinal excitability) will be obtained
Ischemic pain ratings | During PECO and No-PECO conditions (aim #1); Pre-post acute exercise during PECO (aim #2); Pre-post 6 weeks of training during PECO (aim #3)
  Participants will be asked to rate their leg pain intensity twice at the 4-min H-reflex protocol (at 2nd and 4th min of the procedure) using a Cook pain sale (0-10). In the scale, 0 represents no pain while 10 represents the worst possible pain
Arterial blood pressure | During PECO and No-PECO conditions (aim #1); Pre-post acute exercise during PECO (aim #2); Pre-post 6 weeks of training during PECO (aim #3)
  Brachial arterial pressure will be measured twice at the 4-min H-reflex protocol (at 2nd and 4th min of the procedure) by an automated equiment (Tango SunTech Medical)
Pressure pain threshold | Pre-post acute exercise (aim #2); Pre-post 6 weeks of training (aim #3)
  It will be assessed with an analogue algometer (FDK 60, Wagner Instruments) (in rectus femoris, upper-trapezius and biceps brachiis muscles). It measures the kg of force at the time participants report they are feeling pain intead of pressure
Cold pain tolerance | Pre-post acute exercise (aim #2); Pre-post 6 weeks of training (aim #3)
  It will be assessed with participants immersing their right foot into a container with cold water between 0 and 2ºC. It measures the time participants can endure the cold painful stimuli
Cold pain ratings | Pre-post acute exercise (aim #2); Pre-post 6 weeks of training (aim #3)
  While participants immerse their right foot into a container with cold water between 0 and 2ºC, they will beasked to rate the intensity of pain they perceived each minute by writing in a visual analogue scale (0-100mm) that pain intensity. 0 is considered no-pain and 100 the worst possible pain
Heart rate variability during cold pain testing | Pre-post acute exercise (aim #2); Pre-post 6 weeks of training (aim #3)
  It will be measured continuosly during the time participants have their foot in cold water using a heart rate monitor (Polar H10)
Arterial blood pressure during cold pain testing | Pre-post acute exercise (aim #2); Pre-post 6 weeks of training (aim #3)
  It will be measured each minute during the time participants have their foot in cold water using an automatic equipment (Tango SunTech Medical)
Maximal oxygen uptake | Pre-post 6 weeks of training (aim #3)
  For the aerobic group, it will be determined in a treadmill graded exercise testing using a gas analyses system (Metamax, Cortex)
Peak power | Pre-post 6 weeks of training (aim #3)
  For the anaerobic group, it will be determined with a 30-s Wingate all-out test (Monark cycloergometer)
Maximal voluntary isometric contraction | Pre-post 6 weeks of training (aim #3)
  For the dynamic resistance group, it will be determined for the knee extensors muscles using an isokinetic dynamometer (Biodex)
H-reflex after training | Pre-post 6 weeks of training (aim #3)
  With soleus electromyographic recording electrode (Delsys) and electrical stimulation of the tibial nerve (Stimsola) the H-reflex recruitment curve parameters (spinal excitability) will be obtained
V-wave after training | Pre-post 6 weeks of training (aim #3)
  With soleus electromyographic recording electrode (Delsys) and electrical stimulation of the tibial nerve (Stimsola) the V-wave parameters (spinal and supraspinal excitability) will be obtained

CONTACTS AND LOCATIONS:
Overall Officials: Gonçalo V Mendonça, PhD, Principal Investigator — Faculdade de Motricidade Humana
Locations (1):
- Faculdade de Motricidade Humana, Lisbon, Portugal

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT07105410/Prot_SAP_000.pdf